CLINICAL TRIAL: NCT02866461
Title: Endogenous Opioid Systems and Symptom Change in Fibromyalgia
Status: Withdrawn | Type: Observational
Why Stopped: It was not possible to conduct this study at the University of Utah due to the inability of the PET research facility to synthesize the radiotracer central to this project. Project was transferred to another institution.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: R01 3589819
Record Dates: First submitted 2016-03-22; First posted 2016-08-15 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be sampled at baseline to test for genes that may be associated with the function of the chemical signals between nerve cells, function of hormones, and symptoms. The genetic portion of the study is optional.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fibromyalgia: No treatment
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment — Observation

SUMMARY:
This study is designed to study brain mechanisms associated with symptoms and severity of Fibromyalgia. This will be accomplished by relating results from PET scans to self-reported and objective measures of disease severity.

DETAILED DESCRIPTION:
The purpose of this study is to examine µ-opioid receptor (µOR)-mediated neurotransmission in patients diagnosed with persistent pain, fibromyalgia (FM), and its relationship with pain and affect measures. µOR activation is expected to take place in the following brain regions: rostral and dorsal anterior cingulate (rACC, dACC), orbitofrontal cortex (OFC), thalamus (THA), nucleus accumbens (NAC), amygdala (AMY), periaqueductal gray (PAG). Greater regional activation is expected to be associated with improvements in clinical pain ratings and affective state.

The endogenous opioid system and µ-opioid receptors (µORs) play a central role in the regulation of pain, the pathophysiology of chronic pain syndromes, mood and emotion; this system is dysregulated in persistent pain syndromes. A substantial body of literature addressing these mechanisms has been developed in our laboratory, including recent data on the cognitive and molecular mechanisms associated with reductions in pain, as well as trait personality and genetic predictors of emotional effects in the context of pain.

Eighty individuals who have been diagnosed with FM and who fit the inclusion and exclusion criteria will be enrolled in this 14-week protocol. An initial visit for informed consent procedures and baseline characterization will then be scheduled, as well as the visits for positron emission tomography (PET) and magnetic resonance imaging (MRI) procedures. Subjects will return for testing after 6 and 14 weeks.

Volunteers will undergo imaging with structural and functional MRI and PET with [11C]carfentanil to determine baseline µOR non-displaceable binding potential (BPND) and changes in those BPND measures coinciding with symptom severity at the time of scanning.

ELIGIBILITY:
Inclusion Criteria:

* Have met American College of Rheumatology (ACR) criteria for fibromyalgia for at least 1 year;
* Willing to limit introduction of new treatments during the study;
* Use of sleep aids no more than twice per week
* 18-55 years of age
* right handed
* capable of providing written informed consent

Exclusion Criteria:

* concurrent untreated medical illnesses, autoimmune, or inflammatory disease;
* Routine daily use of narcotic analgesics or history of substance abuse;
* Concurrent participation in other therapeutic trials;
* Pregnancy/ nursing;
* Ongoing psychiatric illness;
* Contraindications to PET or MRI methods;
* Impairments that would prevent completion of the study protocol;
* Use of sleep aids at frequency of more that twice per week;
* Allergy to fentanyl

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals diagnosed with Fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
change in mu opioid-mediated neurotransmission | Change from baseline at 6 weeks
  assessed via PET scanning

SECONDARY OUTCOMES:
change in Biomarkers of pain response | Change from baseline at 6 weeks
  serum cortisol
change in Biomarkers of pain response | Change from 8 weeks at 14 weeks
  serum cortisol
change in Pain | Change from baseline at 6 weeks
  assessed via questionnaire
change in Pain | Change from 8 weeks at 14 weeks
  assessed via questionnaire
change in mu opioid-mediated neurotransmission | Change from 8 weeks at 14 weeks
  assessed via PET scanning

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott DJ, Heitzeg MM, Koeppe RA, Stohler CS, Zubieta JK. Variations in the human pain stress experience mediated by ventral and dorsal basal ganglia dopamine activity. J Neurosci. 2006 Oct 18;26(42):10789-95. doi: 10.1523/JNEUROSCI.2577-06.2006. PMID 17050717
- [Background] Harris RE, Clauw DJ, Scott DJ, McLean SA, Gracely RH, Zubieta JK. Decreased central mu-opioid receptor availability in fibromyalgia. J Neurosci. 2007 Sep 12;27(37):10000-6. doi: 10.1523/JNEUROSCI.2849-07.2007. PMID 17855614
- [Background] Harris RE, Zubieta JK, Scott DJ, Napadow V, Gracely RH, Clauw DJ. Traditional Chinese acupuncture and placebo (sham) acupuncture are differentiated by their effects on mu-opioid receptors (MORs). Neuroimage. 2009 Sep;47(3):1077-85. doi: 10.1016/j.neuroimage.2009.05.083. Epub 2009 Jun 6. PMID 19501658
- [Background] Martikainen IK, Pecina M, Love TM, Nuechterlein EB, Cummiford CM, Green CR, Harris RE, Stohler CS, Zubieta JK. Alterations in endogenous opioid functional measures in chronic back pain. J Neurosci. 2013 Sep 11;33(37):14729-37. doi: 10.1523/JNEUROSCI.1400-13.2013. PMID 24027273
- [Background] Pecina M, Martinez-Jauand M, Love T, Heffernan J, Montoya P, Hodgkinson C, Stohler CS, Goldman D, Zubieta JK. Valence-specific effects of BDNF Val66Met polymorphism on dopaminergic stress and reward processing in humans. J Neurosci. 2014 Apr 23;34(17):5874-81. doi: 10.1523/JNEUROSCI.2152-13.2014. PMID 24760847
- [Background] Martikainen IK, Nuechterlein EB, Pecina M, Love TM, Cummiford CM, Green CR, Stohler CS, Zubieta JK. Chronic Back Pain Is Associated with Alterations in Dopamine Neurotransmission in the Ventral Striatum. J Neurosci. 2015 Jul 8;35(27):9957-65. doi: 10.1523/JNEUROSCI.4605-14.2015. PMID 26156996